CLINICAL TRIAL: NCT06534216
Title: Role of Intestinal Ultrasound in Treat to Target Strategy in the Management of Inflammatory Bowel Disease : the IUS-TTT Study
Acronym: IUS-TTT
Status: Active, not recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: Post BH & R 57/03.2024-02
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inflammatory bowel disease: Adult patients with active Inflammatory Bowel Disease (IBD) are eligible for enrollment after obtaining informed consent. Active disease will be defined based on endoscopy with a Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score of 2 or greater for ulcerative colitis, and a Simple Endoscopic Score for Crohn's Disease (SES-CD) of 3 or greater for Crohn's disease.
  Interventions: Diagnostic Test: Intestinal ultrasound

INTERVENTIONS:
Diagnostic Test: Intestinal ultrasound — This study employs intestinal ultrasound (IUS) to assess disease activity in Inflammatory Bowel Disease (IBD) patients. Ultrasound parameters include bowel wall thickness measurement, evaluation of vascularization via color Doppler, assessment of wall stratification, and identification of mesentery features and complications (e.g., strictures, fistulas, abscesses). For ulcerative colitis, disease activity is gauged using the Milan Ultrasound Criteria (MUC), where a score >6.3 indicates active disease based on bowel wall thickness and vascularization. In Crohn's disease, the Bowel Ultrasound Score (BUSS) and International Bowel Ultrasound Segmental Activity Score (IBUS-SAS) assess bowel wall thickness, vascularization, stratification, and inflammatory fat, with scores >3.52 (BUSS) and >48.7 (IBUS-SAS) indicating active disease. IUS evaluations occur at baseline, 2-6 weeks, 12 weeks, and 6-12 months to track disease progression and treatment response.

SUMMARY:
This study aims to evaluate the role of bedside Intestinal Ultrasound (IUS) as a cost-effective, non-invasive, and well-tolerated procedure within the Treat-to-Target strategy for managing Inflammatory Bowel Disease (IBD). Despite its growing use, therapeutic targets for IUS-guided treatment remain inadequately defined. The study will investigate the feasibility of IUS in monitoring transmural response and remission, and its potential to predict clinical and biochemical responses at 3 months, as well as mucosal healing at 6 and 12 months. By incorporating IUS into routine clinical care, we aim to enhance disease management and optimize therapeutic outcomes for patients with ulcerative colitis and Crohn's disease.

DETAILED DESCRIPTION:
This prospective observational pilot study aims to assess the role of Intestinal Ultrasound (IUS) in the management of active Inflammatory Bowel Disease (IBD) over a 6-12 month period at a single tertiary center. The primary objective is to determine the incidence of transmural response at short-term and transmural remission at long-term follow-up. Secondary objectives include evaluating the predictive role of IUS performed at weeks 2-6 for clinical and biochemical response at 3 months, and as a predictor of mucosal healing at 6-12 months. Adult patients with active IBD, defined by endoscopic criteria (Ulcerative Colitis Endoscopic Index of Severity [UCEIS] ≥ 2 for ulcerative colitis and Simple Endoscopic Score for Crohn's Disease [SES-CD] ≥ 3 for Crohn's disease), will be enrolled. Exclusion criteria include age <18 years, Crohn's disease restricted to non-terminal ileum small bowel or gastroduodenal area, normal bowel wall thickness in all segments at week 0, isolated proctitis in ulcerative colitis, body mass index (BMI) >30, and pregnancy. Participants will undergo IUS at baseline, 2-6 weeks, 12 weeks, and 6-12 months, along with measurements of fecal calprotectin, C-reactive protein (CRP), Harvey-Bradshaw Index (HBI), and Simple Clinical Colitis Activity Index (SCCAI), and ileocolonoscopy at baseline and 6-12 months. IUS parameters will include bowel wall thickness, vascularization, wall stratification, mesentery features, and complications. The Milan Ultrasound Criteria (MUC) for ulcerative colitis and the Bowel Ultrasound Score (BUSS) and International Bowel Ultrasound Segmental Activity Score (IBUS-SAS) for Crohn's disease will be used to assess disease activity. Outcomes will measure the incidence of transmural response and remission, and the predictive role of early IUS for clinical, biochemical, and mucosal healing. Ethical clearance is obtained, and informed consent will be taken from all participants. The study aims to enroll 100 patients to gather sufficient data for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years.
* Active Crohn's disease, defined as a Simple Endoscopic Score for Crohn's Disease of 3 or higher.
* Active ulcerative colitis, defined as an Ulcerative Colitis Endoscopic Index of Severity of 2 or higher.

Exclusion Criteria:

* Age < 18 years
* Intestinal ultrasound for assessment of response to therapy
* Intestinal ultrasound for clinically asymptomatic disease
* Pregnancy and lactating mothers

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients with active Inflammatory Bowel Disease (IBD), specifically those diagnosed with either Crohn's disease or ulcerative colitis. To be eligible for enrollment, patients must be over the age of 18 years and must provide informed consent. Active Crohn's disease will be defined as having a Simple Endoscopic Score for Crohn's Disease (SES-CD) of 3 or higher, while active ulcerative colitis will be defined as having an Ulcerative Colitis Endoscopic Index of Severity (UCEIS) of 2 or higher. Patients will be recruited from the Inflammatory Bowel Disease clinic or from inpatients admitted with active disease. Inclusion in the study will only proceed once informed consent has been obtained. This study aims to evaluate the role of intestinal ultrasound in monitoring and guiding the treatment of active IBD, focusing on its feasibility in assessing transmural response and remission as treatment targets.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Change in management | 12 months
  Change in management after intestinal ultrasound as compared to standard of care at different time points (3, 6 and 12 months)

SECONDARY OUTCOMES:
Prediction of clinical and biomarker response | 3 months
  Prediction of clinical and biomarker response at 3 months by 2-6 weeks intestinal ultrasound
Prediction of clinical and biomarker remission | 6 months
  Prediction of clinical and biomarker remission at 6 months by 2-6 weeks and 3 months intestinal ultrasound
Prediction of transmural response | 12 months
  Prediction of transmural response at 3, 6 and 12 months by 2-6 weeks, 3 months and 6 months intestinal ultrasound
Prediction of transmural remission | 12 months
  Prediction of transmural remission at 12 months by 2-6 weeks, 3 months and 6 months intestinal ultrasound
Prediction of endoscopic response and remission | 12 months
  Prediction of endoscopic response and remission at 6-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No